CLINICAL TRIAL: NCT00458952
Title: A Phase I Study Evaluating the Maximum Tolerated Dose, Dosimetry, Safety, and Efficacy of Ultratrace Iobenguane I 131 in Patients With Malignant Pheochromocytoma/Paraganglioma
Brief Title: Phase 1 Study of Iobenguane (MIBG) I 131 in Patients With Malignant Pheochromocytoma/Paraganglioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIP-IB12
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: MIBG; iobenguane; iodine; I 131; radiotherapy; radiopharmaceutical; dosimetry; neuroendocrine tumor; Ultratrace; no carrier added; metaiodobenzyl-guanidine
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Neuroendocrine Tumors | interventions — 3-Iodobenzylguanidine; Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation (Experimental): Dosing of Ultratrace iobenguane I 131 began at 6.0 mCi/kg and escalated in 1.0 mCi/kg increments in order to establish the MTD. The MTD is the dose immediately below the level at which escalation stops due to dose-limiting toxicity (DLT). An additional 3 patients are to be treated at the MTD, for a total of 6.
  Interventions: Drug: Ultratrace Iobenguane (MIBG) I 131

INTERVENTIONS:
Drug: Ultratrace Iobenguane (MIBG) I 131 — Phase I: Dose escalation protocol Phase II: Treatment schedule at therapeutic dose
  Other Names: Ultratrace Iobenguane I 131; Azedra Ultratrace (iobenguane I 131)

SUMMARY:
The purpose of this study is to determine whether iobenguane I 131 is safe and effective in patients with malignant pheochromocytoma or paraganglioma.

DETAILED DESCRIPTION:
This was originally designed as a phase 1/2 study. The phase 1 patients received a small dose of study drug to see if the tumors absorb the drug. If the patient's tumors absorbed the drug, then the patient received one therapeutic dose. In the phase 1 portion, the study employed a 3 + 3 dose escalation design. Enrollment in the phase 1 portion was to be completed once researches believed that they found the highest dose that they could give patients without causing unacceptable toxicity. This dose is called the maximum tolerated dose (MTD). Following discussions with the Food and Drug Administration (FDA) that occurred during the dose escalation stage of the study, the protocol was amended to conclude the trial upon the identification of the MTD. The Phase 2 safety/ efficacy stage of the study was conducted with modifications of the primary endpoint as Protocol MIP IB12B, with Special Protocol Assessment Agreement with the FDA in March 2009.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of either adrenal pheochromocytoma or extra-adrenal paraganglioma by histological confirmation OR plasma-free metanephrines and 24-hour urine test for catecholamines/ metanephrines
* Disease is metastatic or has recurred following surgery
* At least one measurable lesion seen by computed tomography (CT) or magnetic resonance (MR) scan performed within 4 weeks prior to the first dose of study drug
* At least one known tumor site is also seen on Ultratrace iobenguane I 131 scan
* Provide written informed consent and are willing to comply with protocol requirements
* Are at least 18 years of age
* If female, then not of childbearing potential as documented by history (e.g., tubal ligation or hysterectomy) or is post menopausal with a minimum 1 year without menses
* If female of childbearing potential, has a negative serum b-HCG pregnancy test within 48 hours prior to receiving iobenguane I 131
* Females who agree not to become pregnant and males who agree not to father a child during the 1 year period following the therapeutic dose of Ultratrace iobenguane I 131. Both females and males must use an acceptable method of birth control during the first year following the therapeutic dose of Ultratrace iobenguane I 131.

Exclusion Criteria:

* Females who are nursing
* Active CNS lesions by CT/MR scanning within 3 months of study entry
* New York Heart Association class III-IV heart failure
* Received any previous systemic radiotherapy within 6 months of study entry
* Administered prior whole-body radiation therapy
* Received external beam radiotherapy to greater than 25 percent of bone marrow
* Administered prior chemotherapy within 30 days of study entry
* Karnofsky performance status is less than 60
* Platelets are less than 100,000/uL
* Absolute neutrophil count (ANC) is less than 1,500/uL
* Serum creatinine is greater than 1.5 mg/dL
* Total bilirubin is greater than 1.5 times the upper limit of normal
* AST/SGOT or ALT/SGPT is greater than 2.5 times the upper limit of normal
* Has received a therapeutic investigational compound and/or medical device within 30 days before admission into this study
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post dose follow-up examinations
* Is determined by the Investigator that the patient is clinically unsuitable for the study.
* Has received a medication which inhibits uptake of iobenguane I 131:
* phenothiazines or decongestants within 2 weeks prior to enrollment; or,
* a tricyclic antidepressant within 6 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molecular Insight Pharmaceuticals, Study Director — MIP
Locations (3):
- United States (3):
  - New York Presbyterian Hospital-Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Noto RB, Pryma DA, Jensen J, Lin T, Stambler N, Strack T, Wong V, Goldsmith SJ. Phase 1 Study of High-Specific-Activity I-131 MIBG for Metastatic and/or Recurrent Pheochromocytoma or Paraganglioma. J Clin Endocrinol Metab. 2018 Jan 1;103(1):213-220. doi: 10.1210/jc.2017-02030. PMID 29099942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients with confirmed pheochromocytoma/paraganglioma were recruited for participation in the trial at 3 US sites. 21 patients received Ultratrace Iobenguane I 131 while 3 patients failed to meet all inclusion/exclusion criteria and were therefore not dosed.
Pre-assignment Details: Planned Doses: 6, 7, 8 & 9 mCi/kg. Dose reductions in 7, 8 & 9 mCi/kg cohorts were made so total activity administered to pts would not greatly exceed allowed total activity of 525, 600, & 675 mCi for these groups, respectively. Thus, pts were subsequently analyzed in 2 groups of ≤500 mCi and >500mCi, consisting of 7 & 14 patients, respectively.
Groups:
- =< 500 mCi Ultratrace Iobenguane I 131: 7 subjects received a mean dose less than or equal to 500 mCi of Ultratrace Iobenguane I 131
- >500 mCi: 14 subjects received a mean dose of greater than 500 mCi of Ultratrace Iobenguane I 131
Period: Overall Study
Arm/Group | =< 500 mCi Ultratrace Iobenguane I 131 | >500 mCi
Started | 7 | 14
Completed | 5 | 9
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | =< 500 mCi Ultratrace Iobenguane I 131 | >500 mCi | Total
Number analyzed (Participants) | 7 | 14 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 18
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (15.99) | 52.4 (11.41) | 50.4 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 11 | 16
Region of Enrollment [Number; unit: participants]
  United States | 7 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: MTD of Ultratrace Iobenguane I 131
Description: Although no primary efficacy endpoint was defined for this study, the MTD of Ultratrace iobenguane I 131 in patients with malignant pheochromocytoma/paraganglioma (a safety rather than an efficacy parameter) is the primary objective.
Time Frame: 6 weeks post therapy dose
Population: 24 patients with confirmed pheochromocytoma/paraganglioma were recruited for participation in this trial. Of the 24 consenting patients, 21 patients were administered Ultratrace iobenguane I 131. Three patients did not meet all the inclusion and exclusion criteria, and were not allowed into the study.
Measure: Number; unit: mCi/kg
Groups:
- Ultratrace Iobenguane I 131: Each patient was to first receive an imaging dose of 5 mCi of Ultratrace iobenguane I 131 to confirm tumor uptake of the test article. If at least one tumor on a baseline CT/MRI scan was also visualized on the Ultratrace iobenguane I 131 scan, the patient was administered a therapeutic dose of Ultratrace iobenguane I 131. Dosing began at 6 mCi/kg for an initial cohort of 3 patients, and escalated in 1.0 mCi/kg increments until the MTD was established.
Arm/Group | Ultratrace Iobenguane I 131
Number analyzed (Participants) | 21
mCi/kg | 8

ADVERSE EVENTS:
Arm/Group | Ultratrace Iobenguane I 131
Serious Adverse Events (participants affected / at risk) | 15/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultratrace Iobenguane I 131 (N=21)
Chest pain (General disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Spinal disorder (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Thalamic infarction (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1 (2)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ultratrace Iobenguane I 131 (N=21)
Fatigue (General disorders) | 14
Asthenia (General disorders) | 4
Injection site irritation (General disorders) | 3
Edema peripheral (General disorders) | 3
Pyrexia (General disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Anemia (Blood and lymphatic system disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3
Platelet count decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 6
Neutrophil (Investigations) | 5
Blood thyroid stimulating hormone decreased (Investigations) | 4
Hemoglobin decreased (Investigations) | 4
Blood glucose increased (Investigations) | 3
Hematocrit decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 6
Ageusia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less